CLINICAL TRIAL: NCT03756155
Title: The Immediate Effects on Pain Levels After an Isometric Intervention for Individuals With Lateral Elbow Tendinopathy
Brief Title: Isometric Intervention for Lateral Elbow Tendinopathy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI no longer at the institution; departmental permission to deactivate study
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004723
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Lateral Elbow Tendinopathy; Elbow Pain; Elbows Tendonitis; Elbow Sprain; Elbow Injury
MeSH Terms: conditions — Elbow Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two different groups (Group 1 and Group 2) in 10 participant blocks, meaning after every 10 participants eligible and completing the study, there will be 5 participants assigned to each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Group 1 will complete a protocol with 10 sets of 10 second isometric holds followed by 10 second rest intervals between sets. Each repetition will be performed as closely to the targeted 30%-40% value.
  Interventions: Procedure: isometric intervention
- Group 2 (Experimental): Group 2 will complete a protocol with 5 sets of 20 second isometric holds followed by 20 second rest intervals between sets. Each repetition will be performed as closely to the targeted 30% value.
  Interventions: Procedure: isometric intervention

INTERVENTIONS:
Procedure: isometric intervention — The research participants will perform isometric repetitions against the hand held dynamometer
  Other Names: Midrofet hand held dynamometer

SUMMARY:
This study will be looking at people with lateral elbow tendinopathy (elbow pain). The goal is to determine if a one-time isometric intervention will positively change the level of pain and strength as compared to baseline measurements. After determining baseline strength and pain level, an intervention consisting of several trials of isometric hand/wrist contractions will be performed by the participant. Pain and strength will again be assessed immediately after the intervention.

DETAILED DESCRIPTION:
Participants will be randomized into two different groups in 10 participant blocks, meaning after every 10 participants eligible and completing the study, there will be 5 participants assigned to each group. Group 1 will complete a protocol with 10 sets of 10 second isometric holds followed by 10 second rest intervals between sets. Each repetition will be performed as closely to the targeted 30%-40% value. Group 2 will complete a protocol with 5 sets of 20 second isometric holds followed by 20 second rest intervals between sets. Each repetition will be performed as closely to the targeted 30% value. Resistance for both testing conditions will be performed against the examiner's external resistance/against the Microfet hand held dynamometer. Immediately after the intervention, all participants will again repeat their maximal grip on their affected arm using the Jamar hand held dynamometer and will grade their pain level. (The protocol will be identical to the pre testing procedure from above). The pain score and force output will be obtained and documented. Once these steps are complete, testing will cease. All participants will be instructed to follow their referring provider's treatment intervention.

ELIGIBILITY:
Inclusion Criteria:

* - 18 years old or older
* Currently has lateral elbow pain
* If bilateral lateral elbow pain is present, the more symptomatic side will be assessed
* At the time of presentation, individuals have been evaluated as having clinical diagnosed LET for at least 4 weeks
* AND: Positive pain response to at least two of the following tests:

  * Pain with palpation on the affected elbow
  * Pain with resisted wrist or middle finger extension
  * Pain while stretching the lateral forearm muscles (Mills Test)
  * At least 30% deficit of pain-free grip compared with the unaffected side

Exclusion Criteria:

* - Radicular/Cervical conditions reproducing elbow symptoms
* rheumatoid arthritis
* Other elbow pathologies: bursitis, medial epicondylalgia, radial nerve entrapment, posterolateral rotary instability
* History of fracture to the radius, ulna, or humerus with resultant deformity of the involved extremity
* History of an injection within 6 months
* Inability to place the shoulder, elbow and wrist in the required testing position
* The affected elbow had been operated on

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess efficacy: NRS | Randomization through 12 months
  To assess the immediate effects of an isometric intervention on pain levels for individuals with lateral elbow tendinopathy. The primary outcome measure that will be utilized is the Numeric Pain Rating Scale (NRS) which will measure pain intensity using the 11 point scale with values ranging from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Assess correlation between force output during max grip strength testing and reported pain levels | Randomization through 12 months
  To determine if there is a correlation between force output during max grip strength testing and reported pain levels, and to determine if there is a correlation between two different time under tension protocols and max grip strength and reported pain levels. The secondary outcome measure with be grip strength, both pain free and max grip strength which will be measured in pounds using a Jamar handheld dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Chee Vang, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No